CLINICAL TRIAL: NCT02216864
Title: Pilot Split Face Randomized, Evaluator Blinded Study on the Effect of Multiple Subcisions on Rolling Acne Scars
Brief Title: Effect of Multiple Subcisions on Rolling Acne Scars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Professor in Dermatology, Otolaryngology-Head and Neck Surgery, and Surgery, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU97928
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Acne Scars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple Subcision (Experimental): Subjects will receive multiple subcision treatments to their randomized side of the face 5 times total spaced 4 weeks apart.
  Interventions: Procedure: Multiple Subcision
- Control (No Intervention): Subjects will receive no intervention control on the other side of the face.

INTERVENTIONS:
Procedure: Multiple Subcision — At the start of the procedure, a straight vitrectomy knife will be inserted subdermally and will be slowly advanced parallel to the dermis. Rapid advancement and retraction of the needle under the scarred area in a lancing motion will be performed to abrade the underside of the dermis followed by side to side sweeping motions attempting to break any fibrous attachments to the deeper tissues.
  Arms: Multiple Subcision

SUMMARY:
The purpose of this study is to find out whether the use of multiple subcisions over several visits will improve the appearance of rolling acne scars compared to no treatment.

This study was a pilot study designed to determine feasibility of this procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 65
2. Have bilateral rolling acne scars on each side of their face
3. No active or ongoing acne.
4. The subjects are in good health
5. The subject has the willingness and the ability to understand and provide informed consent for the use of their tissue and communicate with the investigator.

Exclusion Criteria:

1. Under 18 years of age
2. Pregnancy or Lactation
3. Subjects who are unable to understand the protocol or to give informed consent
4. Subjects with mental illness
5. Recent Accutane use in the past 6 months
6. Subjects prone to hypertrophic and keloidal scarring
7. Subjects reporting any blood diseases (HIV, Hepatitis, etc.)
8. Subjects reporting a history of Herpes (oral or genital)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-08; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in acne scarring compared to baseline after treatments | Baseline and 36 weeks
  The change in acne scarring is measured using a quantitative global scarring grading system to compare baseline to the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States